CLINICAL TRIAL: NCT06793137
Title: Phase II Trial for Intestinal Microbiome Modulation With Antibiotics in the Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Brief Title: Intestinal Microbiome Modulation With Antibiotics in the Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Samuel Aguiar Jr, MD, PhD, chief of colorectal cancer division at Hospital AC Camargo Cancer Center, AC Camargo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP3589/24
Record Dates: First submitted 2025-01-13; First posted 2025-01-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Rectal Cancer, Adenocarcinoma
Keywords: Total Neoadjuvant Therapy; Intestinal microbiota; Locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Antibiotic in neoadjuvant treatment of locally advanced rectal adenocarcinoma (Experimental): This study investigates the administration of an oral antibiotic, metronidazole, during the first seven days of radiotherapy for patients with locally advanced rectal adenocarcinoma undergoing total neoadjuvant treatment. Metronidazole is a safe medication with a very low risk of adverse effects and is commonly used to treat infections caused by anaerobic bacteria present in the intestinal microbiota. Additionally, certain genera of anaerobic bacteria are known to be associated with a poorer response to treatment.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — This intervention involves administering the oral antibiotic metronidazole during the first seven days of radiotherapy for patients with locally advanced rectal adenocarcinoma who are undergoing total neoadjuvant treatment. Metronidazole is considered a safe medication, with a very low risk of adverse effects. It is commonly used to treat infections caused by anaerobic bacteria that are part of the intestinal microbiota. Additionally, it is well established that certain genera of anaerobic bacteria are linked to a poorer response to treatment.

SUMMARY:
Colorectal cancer is the second most common malignancy worldwide and one-third of these tumors are located in the rectum. The treatment may involve up to three modalities: radiotherapy, chemotherapy, and surgery. For several years, thanks mainly to Brazilian researchers, subgroups of patients have been selected for non-surgical treatment when chemoradiotherapy induces a complete clinical response. These treatment regimens have reached a plateau leading researchers to seek strategies that can increase response rates. Intestinal microbiota studies have shown that an overpopulation of certain anaerobic bacteria is generally associated with poorer treatment response. No study has attempted to intervene in the gut microbiota to increase the complete response rate in rectal cancer. The proposal of the investigators aims to modulate the intestinal microbiota through a phase 2 clinical trial, with the use of metronidazole as the intervention .

DETAILED DESCRIPTION:
This is a single-center, phase 2, single-arm clinical trial, compared with a historical control. The intervention consists of the oral administration of metronidazole at a daily dose of 1.500 mg, divided into three 500mg doses taken every 8 hours, during the first seven days of neoadjuvant radiotherapy. Adherence to metronidazole will be monitored by evaluating records on the patient´s daily card, designed by the researchers, and questioning during medical visits. Adverse events related to metronidazole use are uncommon and mainly include gastrointestinal disturbances. Infrequent reactions occur in less than 0,01% of patients. All adverse effects will be carefully monitored by the study team. Patients may discontinue the medication for any following reasons: disease progression, death, adverse event, leading to permanent discontinuation of chemoradiotherapy, medication intolerance, withdrawal of consent by the patient (or legal representative), or the need for new systemic oncological therapy or surgery. The primary objective of the study is to determine the effectiveness of antimicrobial therapy at the start of neoadjuvant treatment in patients with locally advanced rectal adenocarcinoma. The secondary objectives are to evaluate changes in the intestinal bacterial profile through intestinal analyses (16S RNA analysis) in pre- and post-treatment fecal samples, to measure the organ preservation rate, to determine the rate of complete pathological response among operated patients, to monitor the toxicity of neoadjuvant treatment and to calculate the 3-year locoregional recurrence-free survival rate. The primary outcome will be a complete clinical response to neoadjuvant treatment, defined by the absence of detectable residual disease through the following methods: digital rectal examination, rectal endoscopy, and magnetic resonance image. The standard neoadjuvant treatment regimen consists of long-course radiotherapy, with 4.500 cGy fractionated into 25 applications of 180 cGy, and a boost to the primary tumor up to a total dose of 54 Gy, concomitant with fluoropyrimidine. The current practice is to perform the entire neoadjuvant treatment before surgery, which consists of chemoradiotherapy followed by chemotherapy with fluoropyrimidine and oxaliplatin for up to 6 cycles (TNT consolidation), or starting with chemotherapy followed by chemoradiotherapy (TNT induction). The primary outcome will be evaluated between 7 and 10 days after the completion of chemotherapy in TNT consolidation or between 10-12 weeks after the radiotherapy in TNT induction. For patients who were candidates for rectal amputation and achieved complete clinical response after the neoadjuvant treatment, an organ preservation strategy (Watch Wait - WW) will be recommended as the first option. For patients with mid-rectal tumors, where surgery involves sphincter preservation, total mesorectal excision surgery with sphincter preservation will be offered as the first treatment option, regardless of the response pattern. In cases of complete clinical response, the WW strategy will be offered as an alternative to patients who refuse surgery. For the evaluation of adverse events, patients will be seen before the start of the study, within 7 days of the start of chemoradiotherapy, and at the end of the study, during the evaluation of the primary outcome, with a complete clinical examination and routine laboratory tests. Patients who experience intolerable grade 2 or 3 toxicity will have their treatment dose reduced and/ or interrupted, according to routine procedures. All adverse effects will be graded and assessed to determine if they are treatment-related. Since this is a Brazilian-approved drug that is widely used commercially, the investigators do not expect to observe severe adverse events. However, if there is intolerance, dose reduction will not be allowed, but the investigators will recommend discontinuation. Adverse events will be evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Whenever possible, each adverse event must be evaluated to determine: its severity, its relationship to each study drug, its duration, and actions taken. The investigators will collect pre- and post-intervention stool samples from all patients included in the study to investigate the secondary outcome, which consists of evaluating changes in the intestinal bacteria profile through intestinal analyses (16S RNA analysis) in pre- and post-treatment fecal samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with middle and lower rectal adenocarcinoma, classified as locally advanced or where the tumor´s location necessitates rectal amputation surgery;
* Tumors located below the peritoneal reflection, as determined by MRI, will be defined as middle and lower rectum;
* Patients eligible for rectal amputation will be those with tumor whose distal margin is less than 2,0cm from the pectineal line, as determined by rectoscopy, or less than 2,0cm from the anorectal ring by palpation or MRI.
* Patients with middle rectum cancer candidates for radiotherapy as part of neoadjuvant treatment will be included according to the following criteria: mesorectal fascia compromised by direct extension of the primary tumor or by an affected lymph node; cT4 tumors.

Exclusion Criteria:

* Patients without performance status for total neoadjuvant treatment;
* Histologies other than adenocarcinoma;
* Adenocarcinomas with a microsatellite instability phenotype, as determined by immunohistochemistry;
* Patients with middle rectal tumors who are not indicated for radiotherapy in the neoadjuvant treatment regimen, according to the institutional protocol (tumors cT3N0, with free mesorectal fascia; cT1-3 N+, with free mesorectal fascia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response in total neoadjuvant treatment of rectal adenocarcinoma | Between 7 -10 days after TNT consolidation and 10 - 12 weeks after TNT induction
  Absence of residual disease detectable by clinical examination, rectal endoscopy, nuclear magnetic resonance imaging.

SECONDARY OUTCOMES:
Evaluate changes in the intestinal bacteria profile. | Up to 7 days before starting intervention with metronidazole and up to 7 days after the end of intervention with metronidazole.
  Intestinal analysis (RNA-16S analysis) on fecal samples before and after treatment.
Organ preservation rate. | 6 to 12 weeks after the end of treatment.
  Organ preservation rate after neoadjuvant treatment.
Complete pathological response rate among operated patients | 10 days after surgery.
  Complete pathological response (pCR) in surgical pathological examination result.
Toxicity of neoadjuvant treatment. | Through treatment completion, an average of 6 months.
  Evaluation of neoadjuvant treatment toxicity using CTCAE 5.0.
Locoregional recurrence-free survival. | 3 years after the end of treatment.
  Evaluation of local or locoregional recurrence by magnetic resonance imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Aguiar Jr, MD, PhD, Principal Investigator — A.C. Camargo Cancer Center; Virgilio S Silva, MD, PhD, Study Chair — A.C. Camargo Cancer Center; Renata T Mayumi, MD, Study Chair — A.C. Camargo Cancer Center; Bruna E Catin Kupper, BSN, PhD, Study Chair — A.C. Camargo Cancer Center
Locations (1):
- A.C Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT06793137/Prot_SAP_002.pdf
  • Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT06793137/ICF_003.pdf